CLINICAL TRIAL: NCT01881893
Title: Feasibility Study of the Adult Congenital Heart Disease-Coping and Resilience (ACHD-CARE) Trial
Acronym: ACHD-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOP 123251
Record Dates: First submitted 2013-05-31; First posted 2013-06-20 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Heart Defects, Congenital
Keywords: Quality of life; Psychosocial Support Systems; Randomized Controls as Topic; Cognitive Therapy; Feasibility Studies
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients in this arm of the study will continue to receive their regular level of care.
- ACHD-CARE Program (Experimental): Group based psychosocial intervention.
  * Educational: congenital heart disease information
  * Behavioral: cognitive behavioral therapy
  * Behavioral: social interactions and communication skills
  Interventions: Behavioral: ACHD-CARE Program

INTERVENTIONS:
Behavioral: ACHD-CARE Program — The ACHD-CARE program will be provided in eight 90-minute weekly sessions. The intervention includes information about living with congenital heart disease, cognitive behavioral therapy (CBT) and coping techniques, and opportunities for peer interaction.
  Arms: ACHD-CARE Program

SUMMARY:
The psychosocial development of adults with congenital heart disease (CHD) can be challenged by many issues including family overprotection, impaired peer relationships, delayed progression into independent adulthood, and difficulties with career and future planning. One-third of patients have diagnosable mood or anxiety disorders and the prevalence of depression is 3 times that of the general Canadian population. Unfortunately, most adults with CHD and significant depression or anxiety do not receive mental health treatment. Despite an increasing awareness of the unique psychosocial concerns of this patient population by both health care providers and patients, there have been no interventions targeting psychosocial outcomes in the adult CHD population. Our quantitative and qualitative research suggests that patients themselves are very interested in psychological services that target their distinctive life experiences, are provided in a group setting, and emphasize coping and resilience. The overarching aim of this proposal is to assess the feasibility of a full-scale randomized controlled trial of a group intervention aimed at improving the psychosocial functioning, quality of life, and resilience of adults with CHD.

ELIGIBILITY:
Inclusion Criteria:

* Documented congenital heart disease (CHD), as confirmed by echocardiogram, cardiac catheterization, or previous surgery
* Age greater than or equal to 18 years
* English-language proficiency sufficient to read and complete the consent form and questionnaires and participate in an English-language group
* No planned surgery during patient's participation in the study
* Clinically-elevated score (i.e >=8) on the Hospital Anxiety and Depression Scale depression (HADS-D) or anxiety (HADS-A) subscale

Exclusion Criteria:

* Current psychotherapy or pharmacotherapy
* Significant cognitive impairment, psychosis, or personality disorder as documented in medical chart
* Report of suicidal intent during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Psychosocial Outcome Measures: Change in depression and anxiety symptoms | Prior to randomization (baseline), immediately following the completion of the ACHD-CARE program or Usual Care period, and at three months follow-up
  Symptoms of anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS)

SECONDARY OUTCOMES:
Psychological Outcome Measures: Social functioning | Prior to randomization (baseline), immediately following the completion of the ACHD-CARE program or Usual Care period, and at three months follow-up
  Two metrics will be used to assess social functioning; the Social Functioning subscale of the Short Form Health Status Survey (SF-12v2) and the Enhanced Recovery in Coronary Heart Disease (ENRICHD) Social Support Inventory (ESSI).
Psychosocial Outcome Measures: Resilience | Prior to randomization (baseline), immediately following the completion of the ACHD-CARE program or Usual Care period, and at three months follow-up
  This psychosocial outcome will be measured by the Resilience Scale (RS).
Psychosocial Outcome Measures: Quality of Life and health status | Prior to randomization (baseline), immediately following the completion of the ACHD-CARE program or Usual Care period, and at three months follow-up
  The quality of life of the participants will be measured using the Satisfaction with Life Scales (SWLS) and the Linear Analogue Scale (LAS). Health status will be assessed using the SF-12v2.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne H Kovacs, PhD, Principal Investigator — University Health Network, Toronto; Jane Irvine, PhD, Principal Investigator — University Health Network, York University
Locations (1):
- Toronto Congenital Cardiac Clinic for Adults, Peter Munk Cardiac Centre, Toronto General Hospital, Toronto, Ontario, Canada